CLINICAL TRIAL: NCT02813538
Title: Hypercoagulability and Liver Function After Major Liver Resection
Brief Title: Major Liver Resection: Early Clotting Disorders and Functional Impairment.
Status: Completed | Type: Observational
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Patricia Duque González, MD, PhD, Hospital General Universitario Gregorio Marañon
Other Study IDs: HGUGregorioMaranonCRH2AT
Record Dates: First submitted 2016-06-22; First posted 2016-06-27 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Hepatic Insufficiency; Blood Coagulation Disorders
Keywords: Thrombelastography; Antithrombin proteins; Liver surgery; Liver function tests
MeSH Terms: conditions — Hepatic Insufficiency; Blood Coagulation Disorders | interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Blood samples for anticoagulant proteins levels analysis and thromboelastometry
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IGC and thromboelastometry: Patients that have hyper, normo o hypcoagulability measured by tromboelastometry and anticoagulant proteins levels early after major liver resection and clinical evolution and patients with liver funcion impairment or without it, measured by indocyanine green clearance early after surgery and clinical evolution
  Interventions: Drug: Indocyanine green clearance; Other: Thromboelastometry

INTERVENTIONS:
Drug: Indocyanine green clearance — To evaluate liver function by injection of indocyanine green by a peripheral vein and measure its clearance
  Other Names: Verdye
Other: Thromboelastometry — To evaluate blood coagulation impairment by obtaining blood sample from a peripheral vein and measure anticoagulant proteins levels plus obtaining thromboelastometry

SUMMARY:
The aim of this study is to evaluate early clotting disorders through thromboelastogram and anticoagulant proteins levels (maybe also endothelial markers) and liver function by indocyanine green clearance after major liver resection and search for a potential relationship between them.

DETAILED DESCRIPTION:
We are prospectively recording data from patients undergoing major liver resection. We obtain a full procoagulant and anticoagulant profile preoperatively and, at first, second and sixth day after surgery. We also measure indocyanine green (ICG) clearance preoperatively and in the first two postoperative days. We are also recording clinical data, focusing on medical and surgical complications. We aim to establish the potential value of ICG clearance and or coagulation profile to predict clinical complications

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing major liver surgery defined as resection of 3 or more hepatic segments

Exclusion Criteria:

* Indocyanin green allergy
* Thyrotoxicosis
* Thrombophilia
* Lupus anticoagulant
* Coagulation factor deficiency
* Venous thromboembolism in the last 3 years
* Pulmonary thromboembolism in the last 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major liver surgery defined as resection of 3 or more hepatic segments
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-02-05 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Establish a relationship between ICG and MCF | 1 week
  We aim to find a potential association between ICG and MCF measured by thromboelastometry in the first week after surgery
Establish a relationship between pro and anticoagulant proteins levels and endothelial markers | 1 week
  We aim to find a potential association between procoagulant factor levels, protein C,S and ATIII with thrombomodulin, heparan sulfate and syndecan-1 in the first week after surgery

SECONDARY OUTCOMES:
Study blood coagulation disorders after major liver surgery resection | 2 years
  We aim to characterize blood coagulation disorders during the first week after major liver surgery in our sample of patients
Study liver function after major liver surgery | 2 years
  We aim to study the predictive value of indocyanine green clearance for liver impairment after major liver surgery in our sample of patients

CONTACTS AND LOCATIONS:
Overall Officials: Luis Olmedilla, PhD, Study Director — Gregorio Marañon Hospital
Locations (1):
- Gregorio Marañon Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Publishing results
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From december 2018
Access Criteria: For other researchers and editors